CLINICAL TRIAL: NCT05141383
Title: Comparative Study of Diagnostic and Prognosis Biomarkers of Prostate Cancer in Liquid Biopsy
Brief Title: Comparative Study of Diagnostic and Prognosis Biomarkers of Prostate Cancer in Liquid Biopsy (HOPE)
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2021-04
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer; Healthy Donors
Keywords: diagnostic; prognosis; prostate cancer; long non-coding RNA biomarkers
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 3 cohorts of 118 patients in the aim to have 90 evaluable participants will be included in the study:
  * 40 patients with prostate cancer, or
  * 40 patients with suspected cancer without confirmation on biopsy, or with hyperplasia of the prostate and
  * 38 healthy donors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with prostate cancer (Other): Patients with suspected prostate cancer (MRI or digital rectal examination), or prostatic hyperplasia with a PSA level> 4 ng / ml
  Interventions: Other: Urine sampling
- Patients with suspected cancer without confirmation on biopsy, or with hyperplasia of the prostate (Other): Patients with suspected prostate cancer (MRI or digital rectal examination), or prostatic hyperplasia with a PSA level> 4 ng / ml
  Interventions: Other: Urine sampling
- Healthy donors (Other): Male from 50 to 70 years old with a PSA level <4 ng / mL
  Interventions: Other: Urine sampling

INTERVENTIONS:
Other: Urine sampling — A blood sample and a urine sample after prostate massage will be carried out at baseline
  Other Names: Blood sampling

SUMMARY:
Constitution of a biological collection within the framework of the establishment of a diagnostic, prognostic and active surveillance test for prostate cancer from long non-coding RNA biomarkers, in 3 cohorts of patients, with cancer of the prostate, with suspected cancer without biopsy confirmation or with prostatic hyperplasia and healthy donors.

This biological collection will also be used as a support for further researches on the identification of biomarkers and genetic markers to improve the prognosis and diagnostic management of patients with prostate pathologies.

DETAILED DESCRIPTION:
Multicenter, RIPH 2 study, evaluating on 3 patient cohorts the feasibility of setting up a diagnostic test, prognosis and active surveillance of prostate cancer using long non-coding RNA biomarkers.

For patients agreeing to participate in the study and having signed a consent form, during their routine care consultation in the urology department, will have a blood sample and a urine sample after prostate massage as part of the study, and if necessary, a tissue sample as part of the treatment.

Patients with prostate cancer will be followed as part of their care at least annually, and their follow-up data will be collected as part of the study, without additional sampling.

A blood sample and a urine sample after prostate massage will be carried out during a single consultation at the CIC Henri Mondor for

ELIGIBILITY:
Inclusion Criteria:

Concerning patients:

1. / Patient with suspected prostate cancer or prostatic hyperplasia with a PSA level ≥ 4 ng / ml
2. / Patient diagnosed by prostate MRI in the course of treatment
3. / No infectious episode in the week before the visit (in particular no urinary tract infection) documented by dipstick and absence of fever
4. / Information of the patient and signature of informed consent or his legal representative.
5. / Participant affiliated to a social security scheme

Regarding healthy volunteers:

1. / Male from 50 to 70 years old
2. / PSA level < 4 ng / mL
3. / No infectious episode in the week before the visit (in particular no urinary tract infection), documented by dipstick and the absence of fever
4. / Absence of cancer and history of haematological pathologies < 5 years (in particular leukemia, lymphoma).
5. / Patient information and signature of consent

Exclusion Criteria:

1 / Participants who refused to participate in the biological collection 2) Persons deprived of their liberty or under guardianship. 3) Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer or suspicion of prostate cancer
Enrollment: 80 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Extracting extravesicular particles and RNA from urine fluids | Baseline
  Criteria will be a minimum of 10ng of total RNA extracted per sample total RNA sequencing and greater than 10 million unique reads mapping to the Gencode V32 reference genome.

SECONDARY OUTCOMES:
Extracting extravesicular particles and RNA from blood | Baseline
  Criteria will be a minimum of 10ng of total RNA extracted per sample total RNA sequencing and greater than 10 million unique reads mapping to the Gencode V32 reference genome.

CONTACTS AND LOCATIONS:
Overall Officials: Yves ALLORY, MD PhD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).